CLINICAL TRIAL: NCT02263963
Title: The Transversus Abdominis Plane Block: A Prospective Randomized Clinical Trial Using EXPAREL.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Corewell Health West (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013-066; DDI.FY13.07 (Other: Digestive Disease Institute/Ferguson Clinic)
Record Dates: First submitted 2013-12-02; First posted 2014-10-15 (Estimated); Results first posted 2023-02-28 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-01

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TAP Block Experal (Experimental): Patient who randomized to this arm, will be blinded, TAP block will be performed under ultrasound guidance, where 20-30 ml of Exparel will be injected in transversus abdominis plane, bilaterally.
  Interventions: Drug: Exparel; Procedure: TAP Block
- No TAP Block (No Intervention)

INTERVENTIONS:
Drug: Exparel — In this arm as described above the intervention will be TAP block injection under ultrasound guidance using Exparel.
  Arms: TAP Block Experal
Procedure: TAP Block — no intervention will be done to this arm.
  Arms: TAP Block Experal

SUMMARY:
The purpose of the study is to evaluate the effectiveness of EXPAREL in a transversus abdominis plane block by assessing the demand of postoperative narcotic, length of hospital stay and incidence of postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over the age of 18 years w
2. Elective laparoscopic colorectal resection.

Exclusion Criteria:

1. Patients under 18 years.
2. Patients unable to provide informed consent
3. Patients undergoing emergency surgery.
4. Pregnant women
5. Severe liver or kidney disease (GFR 15-29 ml/min)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-07; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Spectrum Health, Grand Rapids, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- TAP Block Arm: Twenty five patients randomized to this arm. A volume of 7.5 ml of bupivacaine liposome injectable suspension was used for each side of the TAP blocks so that a total of 15 ml were utilized. The remaining 5 ml of bupivacaine liposome injectable suspension were diluted with 30 ml of sterile preservative free saline and used for local infiltration of the laparoscopic wound
- no TAP Block Arm: Twenty five patients randomized to this arm. did not receive TAP block.
Period: Overall Study
Arm/Group | TAP Block Arm | no TAP Block Arm
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- TAP Block: Patient received TAP block
- no TAP Block: patient did not received TAP block
- Total: Total of all reporting groups
Arm/Group | TAP Block | no TAP Block | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 14 | 26
  >=65 years | 13 | 11 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (13.9) | 65.6 (12.5) | 64 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 14 | 25
  Male | 14 | 11 | 25
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Pain Score
Description: Patient will be evaluate for their post operative pain by nurses using visual analog scale from 0 to 10, zero means no pain, 10 is the worst pain can patient ever experience.
Time Frame: participants will be followed for the duration of hospital stay, an expected average of 4 days
Measure: Mean (Full Range); unit: units on a scale
Groups:
- TAP Block: post op pain score
- no TAP Block: postop pain score
Arm/Group | TAP Block | no TAP Block
Number analyzed (Participants) | 25 | 25
units on a scale | 4.2 [0.5 to 8.5] | 4.5 [0 to 9]

2. Secondary Outcome: Postoperative Narcotic Use
Description: Will be measured, by converting all narcotic medicine used during postoperative period to equal morphine in mg, a calculator created by our pharmacy expert is able to convert any narcotic medicine such as fentanyl, oxycodone, hydromorphone, to morphine in mg. By doing that will have one variable to compare to the two groups.
Time Frame: participants will be followed for the duration of hospital stay, an expected average of 4 days
Measure: Mean (Full Range); unit: mg
Groups:
- TAP Block; no TAP Block: post op narcotic use
Arm/Group | TAP Block | no TAP Block
Number analyzed (Participants) | 25 | 25
mg | 85 [0 to 311] | 110 [0 to 461]

3. Other Pre Specified Outcome: Postoperative Complications.
Description: Any postoperative complications within 30 days of procedure, including death will be recorded.
Time Frame: participants will be followed for the duration of hospital stay, and 30 days after discharge.
Measure: Number; unit: participants
Groups:
- TAP Block; no TAP Block: post op ileus
Arm/Group | TAP Block | no TAP Block
Number analyzed (Participants) | 25 | 25
participants | 7 | 9

4. Other Pre Specified Outcome: Length of Hospital Stay.
Description: Length of hospital stay will be measured in number of days patient spends in the hospital from the day of procedure till discharge.
Time Frame: participants will be followed for the duration of hospital stay, an expected average of 4 days
Measure: Mean (Full Range); unit: days
Groups:
- TAP Block; no TAP Block: length of stay
Arm/Group | TAP Block | no TAP Block
Number analyzed (Participants) | 25 | 25
days | 4 [2 to 15] | 4 [2 to 10]

ADVERSE EVENTS:
Groups:
- TAP Block; no TAP Block: adverse event
Arm/Group | TAP Block | no TAP Block
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes